CLINICAL TRIAL: NCT07041372
Title: Cerebral Atherosclerosis Research With Positron Emission Tomography
Acronym: CARPET
Status: Enrolling by invitation | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Min Kim, Professor, Seoul National University Hospital
Other Study IDs: CARPET
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Infarction
Keywords: cerebral infarction
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FDG-PET — The participants undergo whole-body FDG PET once their neurological status has stabilized after stroke.

SUMMARY:
The goal of this clinical trial is to learn if the application of fluorodeoxyglucose positron emission tomography can predict prognosis of stroke patients. The main questions it aims to answer are:

* Does FDG PET can predict future vascular events such as stroke recurrence, myocardial infarction or vascular death among stroke survivors?
* Does FDG PET can predict other important events such as fracture, dementia, bleeding, cancer and overall death among stroke survivors? Researchers will compare the FDG uptake in major organs - such as the amygdala, vertebrae, spleen, liver, internal carotid artery, visceral fat, and psoas muscle - between patients with and without the event of interest to determine whether FDG PET can predict the overall prognosis of stroke patients.

Participants will:

* Undergo whole-body FDG PET once their neurological status has stabilized after stroke.
* Complete questionnaires assessing stress and anxiety (PHQ-9 and PSS-10) on the same day.
* Maintain regular clinic visits for up to 24 months following the index stroke

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke patients who admitted within seven days after symptom onset

Exclusion Criteria:

* Patients with unstable vital signs or neurological symptoms
* Patients with estimated glomerular filtration rate less than 30ml/min
* Patients with uncontrolled diabetes requiring persistent insulin injection
* During pregnancy or while breastfeeding
* Patients with impaired consent capacity
* Patients with diagnosed/treatment for dementia
* Patients undergoing treatment for malignant tumors or serious autoimmune diseases

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 19 years and older who were diagnosed and treated for acute cerebral infarction within 7 days and can voluntarily participate in the study.
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Vascular events | up to 24 months after index stroke
  Stroke, myocardial infarction, vascular death

SECONDARY OUTCOMES:
overall vascular events | up to 24 months after index stroke
  primary vascular events plus transient ischemic attack, venous thromboembolism, peripheral artery disease requiring intervention or hospitalization

OTHER OUTCOMES:
Overall events | up to 24 months after index stroke
  fracture, cancer, bleeding, dementia, overall death

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jong-ro Gu, South Korea

IPD SHARING:
Plan to Share IPD: No